CLINICAL TRIAL: NCT00303264
Title: A Phase II Study to Investigate the Safety and Efficacy of Dexloxiglumide for the Relief of Symptoms of Functional Dyspepsia.
Brief Title: The Safety and Efficacy of Dexloxiglumide for the Relief of Symptoms of Functional Dyspepsia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEX-MD-20
Record Dates: First submitted 2006-03-14; First posted 2006-03-16 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Dyspepsia
Keywords: functional dyspepsia; cholecystokinin; CCK; gastrointestinal; intestinal transit; GI motility; bloating; upper GI discomfort; upper GI; early satiety; nausea; belching; retching; vomiting; GERD
MeSH Terms: conditions — Dyspepsia; Nausea; Eructation; Vomiting; Gastroesophageal Reflux | interventions — dexloxiglumide; Esomeprazole

INTERVENTIONS:
Drug: dexloxiglumide
Drug: Nexium (esomeprazole)

SUMMARY:
"Functional dyspepsia" has been defined loosely as "pain or discomfort centered in the upper abdomen." The symptoms can also include fullness, early satiety, bloating, belching, nausea, retching and vomiting. These symptoms may present with or without the co-existence of symptoms of heartburn or gastroesophageal reflux disease (GERD). Functional dyspepsia is a diagnosis of exclusion in which other disease states, such as ulcer, cancer, etc. are ruled out and the source of the pain is unknown.

The standard of care for most patients presenting with dyspeptic symptoms has been with proton pump inhibitors (PPI), regardless of whether or not the patient's symptoms include acid-related conditions, e.g., heartburn, GERD, etc. Although PPI treatment has yielded some success in these patients, there is a significant population of patients whose dyspeptic symptoms are not adequately treated with PPI's alone.

The purpose of this study is to evaluate the use of dexloxiglumide in the treatment of the symptoms of functional dyspepsia in patients whose dyspeptic symptoms are not being treated adequately with PPI's.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, 18 to 75 years of age, inclusive.
* Must understand English and be able to follow the instructions about completing the diary and questionnaires.
* At the time of Screening, have pain and/or discomfort in your upper abdomen for at least one day each week in the last month.
* At the time of Screening, have at least one other symptom of FD for at least one day each week in the last month.

Exclusion Criteria:

* Have a known hypersensitivity to dexloxiglumide, any PPI, or aluminum/magnesium-containing antacids
* Have a history of organic diseases, structural or biochemical, of the gastrointestinal system that can cause dyspepsia.
* Have active irritable bowel syndrome (C-IBS, alt-IBS, D-IBS).
* Have findings leading to a clinical suspicion of other secondary causes of dyspepsia, including endocrine, metabolic and neurological disorders.
* Have a body mass (BMI) value of greater than 38 (applies to both males and females).
* Have been enrolled in a previous investigational study of dexloxiglumide.
* Have received treatment with any investigational drug within a 30-day period, or 5 half-lives, whichever is longer, prior to study entry.
* Use or dependence on "prohibited" medications at study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in (upper GI) pain/discomfort intensity.

SECONDARY OUTCOMES:
Change from baseline in (upper GI) non-pain symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- For information regarding investigative sites please contact Forest Professional Affairs, St Louis, Missouri, United States